CLINICAL TRIAL: NCT05926869
Title: Comparison of the Efficacy of Clindamycin Phosphate 1% Gel Versus Once-daily Dapsone 5% Gel in the Treatment of Moderate Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Dr. Parisa Sanawar, Principal Investigator, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO.F.2-81/2022-GENL/250/JPMC
Record Dates: First submitted 2023-03-22; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Clindamycin gel (Experimental)
  Interventions: Drug: Clindamycin and Dapsone gel for 03 months
- Group B Dapsone gel (Experimental)
  Interventions: Drug: Clindamycin and Dapsone gel for 03 months

INTERVENTIONS:
Drug: Clindamycin and Dapsone gel for 03 months — Clindamycin is a topical antibiotic which has been widely used in treatment of acne for many decades. Topical Dapsone 5% gel contains sulfone and has an advanced solvent micro particulate delivery system that enables penetration of stratum corneum . It is a new topical drug used in the treatment of Moderate Acne Vulgaris. It has antibacterial as well as anti inflammatory effects

SUMMARY:
Acne vulgaris (AV) is a disease of the pilosebaceous unit that causes noninflammatory lesions (open and closed comedones), inflammatory lesions (papules, pustules, and nodules), and varying degrees of scarring. The key pathogenic processes includes alteration of follicular keratinization that leads to comedones; increased and altered sebum production under androgen control; follicular colonization by Propionibacterium acnes; . The role of topical antibiotics in treating acne is well established. Clindamycin is a topical antibiotic which has been widely used in treatment of acne for many decades. The extensive use of antibiotics in acne has lead to the development of resistance to antimicrobial therapy. Dapsone is known to have antibacterial as well as anti-inflammatory action which may help in reduction of acne.

DETAILED DESCRIPTION:
Topical Dapsone 5% gel contains sulfone and has an advanced solvent micro particulate delivery system that enables penetration of stratum corneum . It is a new topical drug used in the treatment of Moderate Acne Vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* moderate acne vulgaris
* either gender
* 20 to 50 yrs

Exclusion Criteria:

* systemic treatment taken
* pregnant or lactating women
* hematological abnormalities

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the Efficacy of Clindamycin Phosphate 1% Gel Versus Once-daily Dapsone 5% Gel in the Treatment of Moderate Acne Vulgaris | It will be assessed upto 03 months
  Efficacy will be assessed using Global Acne Grading Sore ( GAGS ). For GAGS (Score 1-18 = mild, score 19-30 = moderate, score 31-38 = severe). Mean difference of GAGs score before and after the treatment will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: khadija Asadullah, FCPS, Principal Investigator — Jpmc; Faiza Inam, FCPS, Principal Investigator — Jpmc; Nazia Jabeen, FCPS, Principal Investigator — JPMC
Locations (1):
- JPMC, Karachi, Sindh, Pakistan